CLINICAL TRIAL: NCT02324309
Title: A Single-blind Crossover Study of the Pharmacokinetic and Postprandial Glucose Dynamics of BIOD-531 Compared to Humulin® R U-500 and Humalog® Mix75/25™ in Subjects With Type 2 DM Who Are Treated With ≥ 150 Units of Insulin Per Day
Brief Title: BIOD-531 vs. Humalog Mix 75/25 vs. Humulin R U-500 Post-Meal Glucose Control in Patients With Severe Insulin Resistance
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 3-151
Record Dates: First submitted 2014-12-17; First posted 2014-12-24 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- BIOD-531 pre-meal (Experimental): Subcutaneous injections of 1.2 U/kg before the start of a standardized breakfast and 0.8 U/kg before the start of a standardized dinner.
  Interventions: Drug: BIOD-531
- Humalog Mix 75/25 pre-meal (Active Comparator): Subcutaneous injections of 1.2 U/kg before the start of a standardized breakfast and 0.8 U/kg before the start of a standardized dinner.
  Interventions: Drug: Humalog Mix 75/25
- Humulin R U-500 pre-meal (Active Comparator): Subcutaneous injections of 1.2 U/kg before the start of a standardized breakfast and 0.8 U/kg before the start of a standardized dinner.
  Interventions: Drug: Humulin R U-500
- BIOD-531 post-meal (Experimental): Subcutaneous injections of 1.2 U/kg 20 minutes after the start of a standardized breakfast and 0.8 U/kg 20 minutes after the start of a standardized dinner.
  Interventions: Drug: BIOD-531

INTERVENTIONS:
Drug: BIOD-531
  Arms: BIOD-531 pre-meal
Drug: Humalog Mix 75/25
  Arms: Humalog Mix 75/25 pre-meal
Drug: Humulin R U-500
  Arms: Humulin R U-500 pre-meal
Drug: BIOD-531
  Arms: BIOD-531 post-meal

SUMMARY:
The study is designed to compare meal time glucose control associated with BIOD-531, a rapidly absorbed concentrated insulin to that associated with Humalog Mix 75/25 and Humulin R U-500 in patients with diabetes and severe insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25 kg/m2
* Diabetes Mellitus using ≥ 150 units of insulin or insulin analog per day and/or ≥ 100 units of insulin or insulin analog at a single dosing session for at least 1 month prior to screening
* HbA1c < 10.0%

Exclusion Criteria:

* History of bariatric surgery
* Corticosteroid therapy
* Significant cardiovascular or other major organ disease
* Females who are breast feeding or pregnant
* A sexually active person not using adequate contraceptive methods

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Post-breakfast glucose exposure (AUC) | 0-330 minutes

SECONDARY OUTCOMES:
Speed of insulin absorption (Times to 50%, 90%, maximal insulin concentrations) | 0-330 and 660-1020 minutes
Insulin exposure (AUC) | 0-1440 minutes
Maximal insulin concentration | 0-330 and 660-1020 minutes
Post-lunch and post-dinner glucose exposures (AUC) | 330-660 and 660-1020 minutes
Injection site toleration (VAS and severity scales) | 30 and 690 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Han-Conrad, MD, Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for Clinical Research, Inc. (PICR), Chula Vista, California, United States